CLINICAL TRIAL: NCT03113773
Title: Low Dose Interleukin-2 in Patients With Stable Ischaemic Heart Disease and Acute Coronary Syndromes
Acronym: LILACS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Dr, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LILACS (A093371)
Record Dates: First submitted 2017-03-14; First posted 2017-04-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — aldesleukin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Proleukin/Placebo in patients with stable ischaemic heart disease
  Interventions: Drug: Proleukin; Drug: Placebo Injection
- Part B (Experimental): Proleukin/Placebo in patients with cute coronary syndromes
  Interventions: Drug: Proleukin; Drug: Placebo Injection

INTERVENTIONS:
Drug: Proleukin — Patients will be treated with subcutaneous injections of IL-2 (range 0.3 X 10^6 - 3.0 X 10^6 IU) or placebo once daily for five consecutive days during the trial.A maximum dose of 3.0 X 10^6 IU will be allowed per day.
Drug: Placebo Injection — Dextrose 5%

SUMMARY:
The mainstay for treatment for acute coronary syndrome (ACS) focusses on re-establishing and maintaining the patency of vessels following coronary plaque disruption, through the use of anti-platelets and anticoagulants. Despite advances in management ACS still carries a high risk of morbidity and mortality, thus future management is likely to target other pathways.

Recent studies indicate that CD4+ T cells, and more specifically Treg cells, are important for the control of post-ischemic immune responses and the promotion of myocardial healing. The investigators therefore hypothesise that expansion of Treg cells in patients with ACS dampens the activation of the immune response and promotes both plaque and myocardial healing. The investigators hypothesise that this can be achieved through subcutaneous administration of low doses of interleukin-2 (IL-2). IL-2 supplementation appears to be an attractive therapeutic option playing a key role in Treg cell development, expansion, survival and suppressive function.

DETAILED DESCRIPTION:
This Phase I/II trial will carefully examine the safety of low-dose IL-2 in cardiovascular patients where it is currently contraindicated. The planned doses will be given to the trial patients once a day, over five days as subcutaneous injections [ i) Part A : Repeated doses will be given in the range of 0.3x10^6 IU up to a maximum of 3.0x10^6 IU (total of 25 completed patients across 5 groups: 3:2 randomisation IL-2:placebo) ii) Part B : Repeated doses will be given at doses not exceeding the maximum dose used in Part A (total of 32 completed patients across 4 groups: 6:2 randomisation IL-2:placebo)].

These doses have been chosen on the basis of safety and tolerability data from published clinical studies. In the low dose IL-2 studies evaluated, there were a low rate of adverse events (AEs) in all of the studies with the most commonly reported AEs being injection site reactions, fatigue, fever, nausea and vomiting. A low percentage of serious adverse events (SAEs) were recorded in a GVHD (graft-versus-host disease)-risk study and these SAEs included haemorrhage (CNS), anorexia, and infection (colitis).

The experimental and clinical background in low-dose IL-2 therapy suggests a potential clinical utility of Treg cell expansion in patients with ACS. Administration of low doses of IL-2 in various clinical settings appears to be safe and remarkably efficacious at promoting selective expansion of Treg cells with preserved suppressive function. This is the first trial to assess the mechanism of action of IL-2 therapy in cardiovascular patients. The aim of Part A of this clinical trial is to assess the safety of low-dose IL-2 as well as the proof of mechanism in patients with stable ischaemic heart disease. Part B aims to assess the safety and efficacy of, and increase in Treg as a result of this drug supplementation, in the setting of ACS.

The investigators hypothesize that low doses of IL-2 in patients with ACS can increase Treg number and function, and ultimately promote plaque stabilisation and myocardial healing (this will be further addressed in future studies). In this context, it may improve patient recovery and limit the occurrence/recurrence of major clinical events.

ELIGIBILITY:
Part A

Inclusion Criteria:

* Age 18-75 years old inclusive
* Previous history (≥ 6 months from planned first day of dosing) of coronary artery disease
* No history of recent (< 6 months from planned first day of dosing) admissions for an unstable cardiovascular event e.g. MI (Myocardial Infarction), unstable angina, ACS
* Written informed consent for participation in the trial

Part A

Exclusion Criteria:

* Current presentation with cardiogenic shock (systolic blood pressure <80 mm Hg, unresponsive to fluids, or necessitating catecholamines), severe congestive heart failure and/or pulmonary oedema
* Known active bleeding or bleeding diatheses
* Known active infection requiring antibiotic treatment
* Severe hematologic abnormalities (haematocrit <30% AND platelet cell count of <100 × 10^3/μL AND white blood cell count <3.3 × 10^3/μL )
* Known malignancies requiring active treatment or follow up (However, patients with current/a history of localised basal or squamous cell skin cancer are not excluded from participation in this trial)
* Known heart failure with impaired LV function: echocardiographic findings of LV EF < 45%
* Hypotension (Systolic BP<100mm Hg, DBP<50mmHg) at screening
* Uncontrolled hypertension (>160/100 mmHg) at screening
* History of recurrent syncope (Electrocardiographic history suggestive of arrhythmia syncope (e.g. bifascicular block, sinus bradycardia < 40 beats per minute in absence of sinoatrial block or medications, pre-excited QRS complex, abnormal QT interval, ST segment elevation leads V1 through V3 [Brugada syndrome], negative T wave in right precordial leads and epsilon wave [arrhythmogenic right ventricular dysplasia/cardiomyopathy]))
* Known hepatic failure or abnormal LFTs at baseline (ALT > 2 x ULN).
* Elevated Total Bilirubin Levels, (TBL > 1.5 x ULN) and Alkaline Phosphatase, ALP (ALP > 1.5 x ULN), at baseline
* Acute kidney injury or chronic kidney disease at Stage > 3B (eGFR < 45)
* Respiratory failure
* History of drug induced Stevens Johnson syndrome, Drug reaction with eosinophilia and systemic symptoms (DRESS syndrome), toxic epidermal necrolysis, or contrast allergy (requiring steroid treatment)
* History of recurrent epileptic seizures in the previous 4 years; repetitive or difficult to control seizures, coma or toxic psychosis lasting >48 hours
* If known diabetic, uncontrolled diabetes defined as HbA1c > 64 mmol/mol
* Average corrected QT interval (QTc) > 450 msecs using Bazett's formula using triplicate ECGs (or > 480 msecs if bundle branch block)
* Known chronic active hepatitis (B or C)
* Known HIV infection
* Current infection possibly related to recent or on-going immunosuppressive treatment
* Known autoimmune disease requiring active immunosuppressive therapy
* History of organ transplantation
* Any oral or intravenous Immunosuppressive treatment including Prednisolone, hydrocortisone or disease modifying drugs such as Azathioprine, interferon-alpha, Cyclophosphamide or Mycophenolate. [Other immunosuppressive therapies should be discussed with PI. Inhaled or topical steroids are permissible.]
* Known pregnancy at screening or visit 2 (where applicable)
* On-going lactation
* Inability to comply with trial procedures
* Current participation in the active dosing phase of other interventional clinical trials
* Contra indication to IL-2 treatment or hypersensitivity to IL-2 or to any of its excipients
* Unwillingness or inability to provide written informed consent for participation
* Known hyper- or hypothyroidism
* Any medical history or clinically relevant abnormality that is deemed by the principal investigator/delegate and/or medical monitor to make the patient ineligible for inclusion because of a safety concern

Part B

Inclusion Criteria:

* Age 18-85 years old inclusive
* Current admission (on at least screening visit) with an acute coronary syndrome (non-ST elevation myocardial infarction, i.e., NSTEMI, or unstable angina) with symptoms of myocardial ischemia lasting 10 minutes or more with the patient at rest or with minimal effort plus either elevated levels of TnI on admission or dynamic changes in ECG (new ST-T changes) or T-wave inversion
* Willingness to be dosed within 8 days from initial date of current admission for ACS
* Written informed consent for participation in the trial

Part B

Exclusion Criteria:

* ST elevation myocardial infarction (heart attack) on this admission.
* Current presentation with cardiogenic shock (systolic blood pressure <80 mm Hg, unresponsive to fluids, or necessitating catecholamines), electrical instability, severe congestive heart failure and/or pulmonary oedema
* Known active bleeding or bleeding diatheses
* Known active infection requiring antibiotic treatment
* Severe hematologic abnormalities (haematocrit <30% AND platelet cell count of <100 × 10^3/μL, white blood AND cell count <3.3 × 10^3/μL)
* Known malignancies requiring active treatment or follow up (However, patients with current/a history of localised basal or squamous cell skin cancer are not excluded from participation in this trial)
* Known heart failure with impaired LV function: echocardiographic findings of LV EF < 35%
* Hypotension (Systolic BP (SBP)<100mm Hg, DBP<50mmHg) at screening
* Uncontrolled hypertension (>160/100 mmHg) at screening
* History of recurrent syncope (Electrocardiographic history suggestive of arrhythmia syncope (e.g., bifascicular block, sinus bradycardia < 40 beats per minute in absence of sinoatrial block or medications, pre-excited QRS complex, abnormal QT interval, ST segment elevation leads V1 through V3 [Brugada syndrome], negative T wave in right precordial leads and epsilon wave [arrhythmogenic right ventricular dysplasia/cardiomyopathy]))
* Known hepatic failure or abnormal LFTs at baseline (ALT > 2 x ULN).
* Elevated Total Bilirubin Levels, (TBL > 1.5 x ULN) and Alkaline Phosphatase, ALP (ALP > 1.5 x ULN), at baseline
* Renal impairment at screening (Creatinine clearance [Cockcroft-Gault] <45ml/min)
* Acute respiratory failure
* History of drug induced Stevens Johnson syndrome, Drug reaction with eosinophilia and systemic symptoms (DRESS syndrome), toxic epidermal necrolysis, or contrast allergy (requiring steroid treatment)
* History of recurrent epileptic seizures in the previous 4 years; repetitive or difficult to control seizures, coma or toxic psychosis lasting >48 hours
* Average corrected QT interval (QTc) > 450 msecs using Bazett's formula using triplicate ECGs (or > 480 msecs if bundle branch block)
* Known chronic active hepatitis (B or C)
* Known HIV infection
* Current infection possibly related to recent or on-going immunosuppressive treatment
* Known autoimmune disease requiring active immunosuppressive therapy
* History of organ transplantation
* Any oral or intravenous immunosuppressive treatment including Prednisolone, hydrocortisone or disease modifying drugs such as Azathioprine, interferon-alpha, Cyclophosphamide or Mycophenolate. [Other immunosuppressive therapies should be discussed with PI. Inhaled or topical steroids are permissible.]
* Known pregnancy at screening (where applicable)
* On-going lactation
* Inability to comply with trial procedures
* Current participation in the active dosing phase of other interventional clinical trials
* Contra indication to IL-2 treatment or hypersensitivity to IL-2 or to any of its excipients
* Unwillingness or inability to provide written informed consent for participation
* Known hyper- or hypothyroidism
* Any medical history or clinically relevant abnormality that is deemed by the principal investigator/delegate and/or medical monitor to make the patient ineligible for inclusion because of a safety concern

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Part A - Determination of IL-2 safety and tolerability parameters | Through study completion, average of 24 days
  Biochemistry, haematology, ECGs and adverse events will be reviewed throughout the trial
Part B - Change in the mean circulating Treg levels (percentage of CD4+ T regulatory defined as CD3+, CD4+, CD25high, CD127low cells within the CD3+, CD4+ T cell gate) following treatment with IL-2. | Measured Days 1 and 6
  Percentage change of CD4+ T regulatory cells will be reviewed following treatment with IL-2.
Part B - Determination of IL-2 safety and tolerability parameters | Through study completion, average of 24 days
  Biochemistry, haematology, ECGs and adverse events will be reviewed

SECONDARY OUTCOMES:
Part B - Changes in circulating cardiac biomarkers (including hs-CRP, IL-6, TnI, BNP) | Measured Days 1, 6 and between days 10-24
  Circulating cardiac biomarkers (including hs-CRP, IL-6, TnI, BNP)
Part B - Change in lymphocyte subsets | Measured Days 1 and 6
  Change in lymphocyte subsets
Part B - Pharmacokinetic analysis of IL-2 levels | Measured Days 1 and 6
  PK analysis of IL-2

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBCHB, MA, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao TX, Sriranjan RS, Tuong ZK, Lu Y, Sage AP, Nus M, Hubsch A, Kaloyirou F, Vamvaka E, Helmy J, Kostapanos M, Jalaludeen N, Klatzmann D, Tedgui A, Rudd JHF, Horton SJ, Huntly BJP, Hoole SP, Bond SP, Clatworthy MR, Cheriyan J, Mallat Z. Regulatory T-Cell Response to Low-Dose Interleukin-2 in Ischemic Heart Disease. NEJM Evid. 2022 Jan;1(1):EVIDoa2100009. doi: 10.1056/EVIDoa2100009. Epub 2021 Nov 22. PMID 38319239
- [Derived] Zhao TX, Kostapanos M, Griffiths C, Arbon EL, Hubsch A, Kaloyirou F, Helmy J, Hoole SP, Rudd JHF, Wood G, Burling K, Bond S, Cheriyan J, Mallat Z. Low-dose interleukin-2 in patients with stable ischaemic heart disease and acute coronary syndromes (LILACS): protocol and study rationale for a randomised, double-blind, placebo-controlled, phase I/II clinical trial. BMJ Open. 2018 Sep 17;8(9):e022452. doi: 10.1136/bmjopen-2018-022452. PMID 30224390